CLINICAL TRIAL: NCT00551135
Title: A Randomized, Double Blind Multi Center Dose Ranging Study Of The Efficacy And Safety Of Pregabalin Compared To Placebo In The Adjunctive Treatment Of Post Surgical Pain After Primary Inguinal Hernia Repair
Brief Title: Surgical Pain After Inguinal Hernia Repair (SPAIHR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081171
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Results first posted 2010-07-15 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2010-06

CONDITIONS: Pain, Postoperative; Hernia, Inguinal
Keywords: postoperative pain chronic pain
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 3 (Experimental)
  Interventions: Drug: Pregabalin
- 4 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental)
  Interventions: Drug: Pregabalin
- 1 (Experimental)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — 150 mg BID
  Arms: 3
Drug: placebo — Placebo
  Arms: 4
Drug: Pregabalin — 75 mg BID
  Arms: 2
Drug: Pregabalin — 25 mg BID
  Arms: 1

SUMMARY:
The purpose of this study is to test whether pregabalin added to the standard of care with dosing starting preoperatively and continuing for 1 week post surgery will decrease the intensity of acute post-operative pain following inguinal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* The subject will have elective ( the subject chooses, but does not have to undergo surgery for an emergency) open unilateral inguinal herniorraphy (hernia repair), using mesh Lichtenstein surgery procedure and under general anesthesia and fentanyl or sufentanil/propofol initiation and sevoflurane or isoflurane maintenance plus local anesthetic infiltration at the conclusion of surgery. Study surgery should be anticipated to be in the morning.
* Expected to be able to use and tolerate non-steroidal anti-inflammatory drugs (such as naproxen), tramadol, oxycodone, and acetaminophen/paracetamol for pain control after surgery.
* The subject will be available for a visit within 72 hours of the day of surgery if not admitted the night before for baseline assessments before taking any study medication, and then to receive study medication prior to the day before surgery.
* The subject is expected and agrees to remain at the hospital (or intermediate care facility) for a minimum of 3 hours following surgery.

Exclusion Criteria:

* Subjects with non elective or emergency surgery (must have the surgery no matter what), or hernia with incarceration (the trapping of abdominal contents within the hernia itself).
* Subjects with hernia repair that is not a primary repair. The planned use of nerve block or spinal/epidural/paravertebral anesthesia or surgery is not planned with general anesthesia.
* Subjects that are not allowed to receive the anesthesia agents indicated per protocol and general anesthesia.

Ages: 17 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- United States (19):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, Laguna Hills, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Stony Brook, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Hermitage, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Humble, Texas
  - Pfizer Investigational Site, Kingwood, Texas
- Pfizer Investigational Site, Randwick, New South Wales, Australia
- Canada (3):
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Charlottetown, Prince Edward Island
  - Pfizer Investigational Site, Québec, Quebec
- India (4):
  - Pfizer Investigational Site, Vadodara, Gujarat
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Madurai, Tamil Nadu
  - Pfizer Investigational Site, Delhi
- Spain (3):
  - Pfizer Investigational Site, Alcorcón, Madrid
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
- Sweden (5):
  - Pfizer Investigational Site, Gävle
  - Pfizer Investigational Site, Landskrona
  - Pfizer Investigational Site, Mora
  - Pfizer Investigational Site, Örebro
  - Pfizer Investigational Site, Skellefteå

REFERENCES:
- [Derived] Singla NK, Chelly JE, Lionberger DR, Gimbel J, Sanin L, Sporn J, Yang R, Cheung R, Knapp L, Parsons B. Pregabalin for the treatment of postoperative pain: results from three controlled trials using different surgical models. J Pain Res. 2014 Dec 23;8:9-20. doi: 10.2147/JPR.S67841. eCollection 2015. PMID 25565885
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081171&StudyName=Surgical%20Pain%20After%20Inguinal%20Hernia%20Repair%20%28SPAIHR%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male subjects were enrolled at 34 centers and participated in the study between 18 January 2008 and 14 September 2009.
Groups:
- Pregabalin 50 mg: Pregabalin 25 milligrams (mg) administered orally (PO) the evening before surgery and 2+/-1 hours before surgery, then Pregabalin 25 mg twice daily (BID) PO for 1 week until Day 7 post surgery (End of Treatment or Beginning of Taper visit), followed by Placebo 25 mg PO BID for 1 week.
- Pregabalin 150 mg: Pregabalin 75 mg administered PO the evening before surgery and 2+/-1 hours before surgery, then Pregabalin 75 mg BID PO for 1 week until Day 7 post surgery (End of Treatment or Beginning of Taper visit), followed by Placebo 75 mg PO BID for 1 week.
- Pregabalin 300 mg: Pregabalin 150 mg administered PO the evening before surgery and 2+/-1 hours before surgery, then Pregabalin 150 mg BID PO for 1 week until Day 7 post surgery (End of Treatment or Beginning of Taper visit), followed by Placebo 150 mg PO BID for 1 week.
- Placebo: Placebo capsules administered PO the evening before surgery and 2+/-1 hours before surgery, then Placebo capsules BID PO for 1 week until Day 7 post surgery (End of Treatment or Beginning of Taper visit), followed by Placebo capsules BID for 1 week.
Period: Overall Study
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Started | 108 | 106 | 103 | 108
Completed | 103 | 104 | 98 | 103
Not Completed | 5 | 2 | 5 | 5
Not completed — Adverse Event | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Other | 3 | 2 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo | Total
Number analyzed (Participants) | 108 | 106 | 103 | 108 | 425
Age, Customized [Number; unit: participants]
  Between 18 and 44 years | 43 | 37 | 40 | 46 | 166
  Between 45 and 64 years | 48 | 58 | 52 | 47 | 205
  >=65 years | 17 | 11 | 11 | 15 | 54
Sex/Gender, Customized [Number; unit: participants] — Number of male subjects
  participants | 108 | 106 | 103 | 108 | 425

OUTCOME MEASURES:

1. Primary Outcome: Modified Brief Pain Inventory-Short Form (mBPI-sf): Worst Pain 24 Hours Post Surgery
Description: m-BPI-sf: a self-administered 11-point Likert rating scale to rate pain in the past 24 hours. A single item pertains to worst pain in the past 24 hours: range of 0 (no pain) to 10 (worst imaginable pain).
Time Frame: 24 hours post surgery
Population: Modified Intent-to-Treat Population (MITT): all subjects included in intent-to-treat population who took study medication 12 and 2 hours prior to surgery, had no complications during herniorrhaphy, and had the post-surgery primary efficacy measurement. Data from 1 site excluded due to Good Clinical Practices (GCP) deviations.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on scale | 5.2 (0.24) | 5.4 (0.25) | 4.7 (0.24) | 5.4 (0.24)
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; LS Means from ANOVA model with terms of treatment, pooled center and baseline worst pain (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0668, ANOVA — Hochberg's adjustment applied to p-value; Hochberg's adjusted p-value was the primary analysis
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; LS (least squares) means from ANOVA model with terms of treatment, pooled center and baseline worst pain (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0334, ANOVA — Unadjusted (raw) p-value
Statistical Analysis 3: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8003, ANOVA — Hochberg's adjustment applied to p-value; Hochberg's adjusted p-value was the primary analysis
Statistical Analysis 4: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8003, ANOVA — Unadjusted (raw) p-value
Statistical Analysis 5: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6932, ANOVA — Unadjusted (raw) p-value

2. Secondary Outcome: Numeric Rating Scale (NRS): Current Pain With Movement - Sitting
Description: NRS: a self-administered questionnaire to rate pain. A single item asks to rate pain with movement caused by sitting (sitting in a standardized fashion after being in a fully supine position); range: 0 (no pain) to 10 (worst pain).
Time Frame: Baseline; 2 hours (h) before surgery (BS); 1, 2, and 3 h post surgery (PS); Days 2, 3, 4, 5, 6, and 7 PS; and End of Treatment (EOT [Day 7 PS or Early Termination])
Population: MITT; data from 1 site excluded due to GCP deviations; n=number of subjects with analyzable data at observation (pregabalin 50 mg, pregabalin 150 mg, pregabalin 300 mg, and placebo, respectively).
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on scale
  Baseline | 1.3 (0.17) | 1.2 (0.18) | 1.0 (0.17) | 1.1 (0.17)
  2 h BS (n=102, 99, 101, 101) | 0.7 (0.10) | 0.6 (0.10) | 0.8 (0.10) | 0.9 (0.10)
  1 h PS (n=92, 91, 91, 91) | 3.6 (0.24) | 4.1 (0.24) | 3.1 (0.24) | 4.1 (0.24)
  2 h PS (n=96, 93, 100, 96) | 3.3 (0.21) | 3.7 (0.21) | 3.2 (0.20) | 3.5 (0.21)
  3 h PS (n=100, 98, 101, 101) | 2.7 (0.19) | 3.3 (0.19) | 2.9 (0.18) | 3.1 (0.19)
  Day 2 PS (n=102, 98, 101, 100) | 3.5 (0.22) | 3.6 (0.23) | 3.4 (0.22) | 3.7 (0.22)
  Day 3 PS (n=102, 98, 100, 101) | 2.7 (0.22) | 3.0 (0.22) | 3.0 (0.22) | 2.8 (0.22)
  Day 4 PS (n=101, 99, 99, 101) | 2.2 (0.20) | 2.2 (0.20) | 2.4 (0.20) | 2.3 (0.20)
  Day 5 PS (n=101, 99, 98, 100) | 1.7 (0.18) | 1.8 (0.18) | 1.9 (0.18) | 2.0 (0.18)
  Day 6 PS (n=100, 99, 98, 99) | 1.6 (0.17) | 1.6 (0.17) | 1.8 (0.17) | 1.7 (0.17)
  Day 7 PS (n=96, 93, 91, 93) | 1.5 (0.17) | 1.5 (0.17) | 1.8 (0.18) | 1.5 (0.17)
  EOT (n=101, 99, 100, 100) | 1.0 (0.15) | 1.3 (0.15) | 1.3 (0.15) | 1.2 (0.15)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; Baseline; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from sitting (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.4471, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7248, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7556, ANOVA
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; 2 h BS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from sitting (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0571, ANOVA
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0197, ANOVA
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.2398, ANOVA
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; 1 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from sitting (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0709, ANOVA
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.9902, ANOVA
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.0018, ANOVA
Statistical Analysis 10: Comparison: Pregabalin 50 mg vs Placebo; 2 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from sitting (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.4639, ANOVA
Statistical Analysis 11: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; p = 0.4845, ANOVA
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; p = 0.1641, ANOVA
Statistical Analysis 13: Comparison: Pregabalin 50 mg vs Placebo; 3 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from sitting (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.1025, ANOVA
Statistical Analysis 14: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.5615, ANOVA
Statistical Analysis 15: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.2904, ANOVA
Statistical Analysis 16: Comparison: Pregabalin 50 mg vs Placebo; Day 2 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from sitting (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.6017, ANOVA
Statistical Analysis 17: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; p = 0.8549, ANOVA
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; p = 0.3386, ANOVA
Statistical Analysis 19: Comparison: Pregabalin 50 mg vs Placebo; Day 3 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from sitting (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.7070, ANOVA
Statistical Analysis 20: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 2, analysis 19]; Test type: Superiority or Other; p = 0.5244, ANOVA
Statistical Analysis 21: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 2, analysis 19]; Test type: Superiority or Other; p = 0.4245, ANOVA
Statistical Analysis 22: Comparison: Pregabalin 50 mg vs Placebo; Day 4 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from sitting (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.8624, ANOVA
Statistical Analysis 23: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 2, analysis 22]; Test type: Superiority or Other; p = 0.7552, ANOVA
Statistical Analysis 24: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 2, analysis 22]; Test type: Superiority or Other; p = 0.7329, ANOVA
Statistical Analysis 25: Comparison: Pregabalin 50 mg vs Placebo; Day 5 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from sitting (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.3053, ANOVA
Statistical Analysis 26: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 2, analysis 25]; Test type: Superiority or Other; p = 0.5290, ANOVA
Statistical Analysis 27: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 2, analysis 25]; Test type: Superiority or Other; p = 0.7951, ANOVA
Statistical Analysis 28: Comparison: Pregabalin 50 mg vs Placebo; Day 6 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from sitting (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.7150, ANOVA
Statistical Analysis 29: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 2, analysis 28]; Test type: Superiority or Other; p = 0.4566, ANOVA
Statistical Analysis 30: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 2, analysis 28]; Test type: Superiority or Other; p = 0.7750, ANOVA
Statistical Analysis 31: Comparison: Pregabalin 50 mg vs Placebo; Day 7 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from sitting (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.9241, ANOVA
Statistical Analysis 32: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 2, analysis 31]; Test type: Superiority or Other; p = 0.8994, ANOVA
Statistical Analysis 33: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 2, analysis 31]; Test type: Superiority or Other; p = 0.2088, ANOVA
Statistical Analysis 34: Comparison: Pregabalin 50 mg vs Placebo; EOT; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from sitting (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2152, ANOVA
Statistical Analysis 35: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 2, analysis 34]; Test type: Superiority or Other; p = 0.7662, ANOVA
Statistical Analysis 36: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 2, analysis 34]; Test type: Superiority or Other; p = 0.7579, ANOVA

3. Secondary Outcome: Numeric Rating Scale (NRS): Current Pain With Movement - Walking
Description: NRS: a self-administered questionnaire to rate pain. A single item asks to rate pain with movement caused by walking (rising from sitting position and walking approximately 5 meters or 16 feet at a moderate pace); range: 0 (no pain) to 10 (worst pain).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on scale
  Baseline | 1.9 (0.23) | 1.6 (0.24) | 1.9 (0.23) | 2.0 (0.23)
  2 h BS (n=102, 98, 101, 101) | 1.2 (0.12) | 1.1 (0.12) | 1.2 (0.12) | 1.2 (0.12)
  1 h PS (n=69, 62, 63, 60) | 3.2 (0.29) | 3.9 (0.32) | 2.9 (0.31) | 3.7 (0.32)
  2 h PS (n=84, 76, 84, 80) | 3.3 (0.27) | 3.4 (0.28) | 3.1 (0.25) | 3.6 (0.27)
  3 h PS (n=96, 91, 93, 94) | 3.1 (0.22) | 3.6 (0.23) | 3.0 (0.22) | 3.3 (0.23)
  Day 2 PS (n=102, 98, 101, 100) | 3.3 (0.23) | 3.8 (0.23) | 3.3 (0.23) | 3.9 (0.23)
  Day 3 PS (n=102, 98, 100, 101) | 2.7 (0.21) | 3.0 (0.22) | 2.8 (0.21) | 2.9 (0.21)
  Day 4 PS (n=101, 99, 99, 101) | 2.2 (0.20) | 2.2 (0.20) | 2.1 (0.20) | 2.2 (0.20)
  Day 5 PS (n=101, 99, 98, 100) | 1.7 (0.17) | 1.8 (0.17) | 1.8 (0.17) | 1.9 (0.17)
  Day 6 PS (n=100, 99, 98, 99) | 1.5 (0.17) | 1.6 (0.17) | 1.7 (0.17) | 1.6 (0.17)
  Day 7 PS (n=96, 93, 91, 93) | 1.3 (0.17) | 1.4 (0.17) | 1.5 (0.17) | 1.3 (0.17)
  EOT (n=101, 99, 100, 100) | 1.1 (0.16) | 1.2 (0.16) | 1.3 (0.16) | 1.2 (0.16)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; Baseline; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from walking (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.6896, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1934, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.6034, ANOVA
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; 2 h BS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from walking (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.7992, ANOVA
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.4770, ANOVA
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.8730, ANOVA
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; 1 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from walking (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2000, ANOVA
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.5059, ANOVA
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.0348, ANOVA
Statistical Analysis 10: Comparison: Pregabalin 50 mg vs Placebo; 2 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from walking (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.3815, ANOVA
Statistical Analysis 11: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 3, analysis 10]; Test type: Superiority or Other; p = 0.4716, ANOVA
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 3, analysis 10]; Test type: Superiority or Other; p = 0.1063, ANOVA
Statistical Analysis 13: Comparison: Pregabalin 50 mg vs Placebo; 3 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from walking (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.3884, ANOVA
Statistical Analysis 14: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; p = 0.3787, ANOVA
Statistical Analysis 15: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; p = 0.2537, ANOVA
Statistical Analysis 16: Comparison: Pregabalin 50 mg vs Placebo; Day 2 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from walking (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0952, ANOVA
Statistical Analysis 17: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.7725, ANOVA
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.0660, ANOVA
Statistical Analysis 19: Comparison: Pregabalin 50 mg vs Placebo; Day 3 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from walking (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.3657, ANOVA
Statistical Analysis 20: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 3, analysis 19]; Test type: Superiority or Other; p = 0.7717, ANOVA
Statistical Analysis 21: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 3, analysis 19]; Test type: Superiority or Other; p = 0.5849, ANOVA
Statistical Analysis 22: Comparison: Pregabalin 50 mg vs Placebo; Day 4 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from walking (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.9580, ANOVA
Statistical Analysis 23: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 3, analysis 22]; Test type: Superiority or Other; p = 0.9884, ANOVA
Statistical Analysis 24: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 3, analysis 22]; Test type: Superiority or Other; p = 0.6743, ANOVA
Statistical Analysis 25: Comparison: Pregabalin 50 mg vs Placebo; Day 5 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from walking (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2689, ANOVA
Statistical Analysis 26: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; p = 0.6907, ANOVA
Statistical Analysis 27: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; p = 0.4798, ANOVA
Statistical Analysis 28: Comparison: Pregabalin 50 mg vs Placebo; Day 6 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from walking (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.5609, ANOVA
Statistical Analysis 29: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 3, analysis 28]; Test type: Superiority or Other; p = 0.9834, ANOVA
Statistical Analysis 30: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 3, analysis 28]; Test type: Superiority or Other; p = 0.8339, ANOVA
Statistical Analysis 31: Comparison: Pregabalin 50 mg vs Placebo; Day 7 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from walking (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.8730, ANOVA
Statistical Analysis 32: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 3, analysis 31]; Test type: Superiority or Other; p = 0.6327, ANOVA
Statistical Analysis 33: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 3, analysis 31]; Test type: Superiority or Other; p = 0.3986, ANOVA
Statistical Analysis 34: Comparison: Pregabalin 50 mg vs Placebo; EOT; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from walking (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.6370, ANOVA
Statistical Analysis 35: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 3, analysis 34]; Test type: Superiority or Other; p = 0.9869, ANOVA
Statistical Analysis 36: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 3, analysis 34]; Test type: Superiority or Other; p = 0.7550, ANOVA

4. Secondary Outcome: Numeric Rating Scale (NRS): Current Pain With Movement - Coughing
Description: NRS: a self-administered questionnaire to rate pain. A single item asks to rate pain with movement caused by coughing (coughing two times while sitting); range: 0 (no pain) to 10 (worst pain)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on scale
  Baseline | 2.4 (0.25) | 1.8 (0.26) | 2.2 (0.26) | 2.1 (0.26)
  2 h BS (n=102, 99, 101, 101) | 1.4 (0.15) | 1.5 (0.15) | 1.6 (0.15) | 1.8 (0.15)
  1 h PS (n=95, 91, 93, 90) | 4.4 (0.26) | 4.8 (0.26) | 3.7 (0.26) | 4.6 (0.26)
  2 h PS (n=96, 93, 99, 97) | 4.1 (0.23) | 4.3 (0.24) | 3.8 (0.23) | 4.3 (0.23)
  3 h PS (n=100, 99, 100, 100) | 3.8 (0.22) | 4.1 (0.22) | 3.8 (0.22) | 3.9 (0.22)
  Day 2 PS (n=102, 98, 101, 100) | 4.6 (0.25) | 5.1 (0.26) | 4.5 (0.25) | 5.2 (0.25)
  Day 3 PS (n=102, 98, 101, 100) | 4.3 (0.24) | 4.5 (0.25) | 4.3 (0.25) | 4.5 (0.24)
  Day 4 PS (n=101, 99, 99, 101) | 3.6 (0.25) | 3.6 (0.25) | 3.6 (0.25) | 3.9 (0.25)
  Day 5 PS (n=101, 99, 98, 100) | 2.8 (0.24) | 3.1 (0.24) | 3.2 (0.24) | 3.8 (0.24)
  Day 6 PS (n=100, 99, 98, 99) | 2.6 (0.23) | 2.8 (0.23) | 2.9 (0.23) | 3.2 (0.23)
  Day 7 PS (n=96, 93, 91, 93) | 2.4 (0.23) | 2.5 (0.24) | 2.5 (0.24) | 2.7 (0.23)
  EOT (n=101, 99, 100, 100) | 1.9 (0.21) | 2.0 (0.21) | 2.3 (0.21) | 2.3 (0.21)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; Baseline; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from coughing (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2912, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.3723, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.6116, ANOVA
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; 2 h BS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from coughing (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0835, ANOVA
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.1497, ANOVA
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.3950, ANOVA
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; 1 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from coughing (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.5892, ANOVA
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.6143, ANOVA
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.0104, ANOVA
Statistical Analysis 10: Comparison: Pregabalin 50 mg vs Placebo; 2 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from coughing (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.5666, ANOVA
Statistical Analysis 11: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p = 0.9008, ANOVA
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p = 0.0967, ANOVA
Statistical Analysis 13: Comparison: Pregabalin 50 mg vs Placebo; 3 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from coughing (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.8353, ANOVA
Statistical Analysis 14: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.4530, ANOVA
Statistical Analysis 15: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.7297, ANOVA
Statistical Analysis 16: Comparison: Pregabalin 50 mg vs Placebo; Day 2 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from coughing (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0692, ANOVA
Statistical Analysis 17: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.6333, ANOVA
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.0325, ANOVA
Statistical Analysis 19: Comparison: Pregabalin 50 mg vs Placebo; Day 3 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from coughing (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.5788, ANOVA
Statistical Analysis 20: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; p = 0.9224, ANOVA
Statistical Analysis 21: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; p = 0.5527, ANOVA
Statistical Analysis 22: Comparison: Pregabalin 50 mg vs Placebo; Day 4 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from coughing (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2624, ANOVA
Statistical Analysis 23: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p = 0.3263, ANOVA
Statistical Analysis 24: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p = 0.3746, ANOVA
Statistical Analysis 25: Comparison: Pregabalin 50 mg vs Placebo; Day 5 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from coughing (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0050, ANOVA
Statistical Analysis 26: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 4, analysis 25]; Test type: Superiority or Other; p = 0.0493, ANOVA
Statistical Analysis 27: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 4, analysis 25]; Test type: Superiority or Other; p = 0.0773, ANOVA
Statistical Analysis 28: Comparison: Pregabalin 50 mg vs Placebo; Day 6 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from coughing (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0547, ANOVA
Statistical Analysis 29: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 4, analysis 28]; Test type: Superiority or Other; p = 0.1976, ANOVA
Statistical Analysis 30: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 4, analysis 28]; Test type: Superiority or Other; p = 0.3832, ANOVA
Statistical Analysis 31: Comparison: Pregabalin 50 mg vs Placebo; Day 7 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from coughing (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.4216, ANOVA
Statistical Analysis 32: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 4, analysis 31]; Test type: Superiority or Other; p = 0.5852, ANOVA
Statistical Analysis 33: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 4, analysis 31]; Test type: Superiority or Other; p = 0.7336, ANOVA
Statistical Analysis 34: Comparison: Pregabalin 50 mg vs Placebo; EOT; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain from coughing (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.1647, ANOVA
Statistical Analysis 35: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 4, analysis 34]; Test type: Superiority or Other; p = 0.2813, ANOVA
Statistical Analysis 36: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 4, analysis 34]; Test type: Superiority or Other; p = 0.8423, ANOVA

5. Secondary Outcome: Numeric Rating Scale (NRS): Current Pain With Movement - Area Under the Curve (AUC) for Sitting, Walking, and Coughing
Description: NRS: a self-administered questionnaire to rate pain. AUC from 1 h PS through 48 h PS for ratings of pain caused by movements of sitting, walking, and coughing; Range: 0 (no pain) to 10 (worst pain).
Time Frame: 1 hour through 48 hours post surgery
Population: MITT; 1 site excluded for GCP deviations; n=subjects with analyzable data at observation (pregabalin 50, 150, and 300 mg, and placebo, respectively).
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on scale
  Sitting (n=100, 99, 101, 101) | 146.22 (8.185) | 158.90 (8.261) | 148.25 (8.115) | 155.57 (8.125)
  Walking (n=97, 91, 95, 96) | 143.82 (8.981) | 162.70 (9.575) | 143.40 (9.063) | 161.74 (9.235)
  Coughing (n=101, 99, 100, 101) | 202.93 (9.635) | 219.69 (9.778) | 199.13 (9.645) | 220.34 (9.601)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; Sitting; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain caused by sitting. Centers with fewer than 8 treated subjects were combined into pooled centers. Last observation carried forward algorithm or first non-missing observation carried backward algorithm applied to missing scores 1-3 h PS and independently to missing scores 24-48 h PS, before applying trapezoidal rule to compute AUC. AUC=missing if all scores 1-3 or 24-48 h PS missing; Test type: Superiority or Other; p = 0.3970, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.7640, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.5064, ANOVA
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; Walking; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain caused by walking. Centers with fewer than 8 treated subjects were combined into pooled centers. Last observation carried forward algorithm or first non-missing observation carried backward algorithm applied to missing scores 1-3 h PS and independently to missing scores 24-48 h PS, before applying trapezoidal rule to compute AUC. AUC=missing if all scores 1-3 or 24-48 h PS missing; Test type: Superiority or Other; p = 0.1318, ANOVA
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; p = 0.9367, ANOVA
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; p = 0.1259, ANOVA
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; Coughing; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain caused by coughing. Centers with fewer than 8 treated subjects were combined into pooled centers. Last observation carried forward algorithm or first non-missing observation carried backward algorithm applied to missing scores 1-3 h PS and independently to missing scores 24-48 h PS, before applying trapezoidal rule to compute AUC. AUC=missing if all scores 1-3 or 24-48 h PS missing; Test type: Superiority or Other; p = 0.1812, ANOVA
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.9600, ANOVA
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.1050, ANOVA

6. Secondary Outcome: Numerical Rating Scale (NRS): Current Pain at Rest
Description: NRS: a self-administered questionnaire to rate pain. A single item asks participant to rate current pain at rest (preceding pain with movement); range: 0 (no pain) to 10 (worst pain).
Time Frame: 2 hours (h) before surgery (BS); 1, 2, and 3 h post surgery (PS); Days 2, 3, 4, 5, 6, 7, 8, 9, and 10 PS
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on scale
  2 h BS (n=102, 99, 101, 101) | 0.9 (0.11) | 0.7 (0.12) | 0.8 (0.11) | 0.7 (0.11)
  1 h PS (n=102, 97, 100, 100) | 3.3 (0.20) | 3.7 (0.20) | 2.9 (0.20) | 3.8 (0.20)
  2 h PS (n=102, 99, 101, 101) | 3.1 (0.18) | 3.2 (0.18) | 2.7 (0.18) | 3.0 (0.18)
  3 h PS (n=102, 99, 101, 101) | 2.5 (0.17) | 2.7 (0.18) | 2.6 (0.17) | 2.7 (0.17)
  Day 2 PS (n=101, 99, 100, 101) | 3.2 (0.22) | 3.3 (0.23) | 3.3 (0.22) | 3.3 (0.22)
  Day 3 PS (n=102, 99, 100, 100) | 2.5 (0.19) | 2.7 (0.19) | 2.2 (0.19) | 2.3 (0.19)
  Day 4 PS (n=101, 99, 99, 101) | 2.0 (0.18) | 2.0 (0.18) | 1.9 (0.18) | 1.8 (0.18)
  Day 5 PS (n=101, 98, 98, 100) | 1.4 (0.17) | 1.8 (0.17) | 1.8 (0.17) | 1.7 (0.17)
  Day 6 PS (n=100, 99, 98, 98) | 1.3 (0.15) | 1.4 (0.15) | 1.4 (0.15) | 1.5 (0.15)
  Day 7 PS (n=96, 93, 90, 93) | 1.2 (0.14) | 1.4 (0.14) | 1.3 (0.14) | 1.3 (0.14)
  Day 8 PS (n=60, 62, 53, 60) | 1.3 (0.19) | 1.2 (0.19) | 1.2 (0.20) | 1.1 (0.19)
  Day 9 PS (n=21, 24, 25, 22) | 0.4 (0.21) | 1.0 (0.20) | 0.6 (0.20) | 1.5 (0.19)
  Day 10 PS (n=11, 11, 13, 11) | 0.5 (0.33) | 1.0 (0.33) | 0.9 (0.31) | 0.9 (0.29)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; 2 h BS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2818, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.8631, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.5074, ANOVA
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; 1 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0401, ANOVA
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.5509, ANOVA
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.0004, ANOVA
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; 2 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.7070, ANOVA
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.3840, ANOVA
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.2732, ANOVA
Statistical Analysis 10: Comparison: Pregabalin 50 mg vs Placebo; 3 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.4418, ANOVA
Statistical Analysis 11: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.8379, ANOVA
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.5944, ANOVA
Statistical Analysis 13: Comparison: Pregabalin 50 mg vs Placebo; Day 2 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.8139, ANOVA
Statistical Analysis 14: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.9709, ANOVA
Statistical Analysis 15: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.9666, ANOVA
Statistical Analysis 16: Comparison: Pregabalin 50 mg vs Placebo; Day 3 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.3204, ANOVA
Statistical Analysis 17: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 16]; Test type: Superiority or Other; p = 0.0869, ANOVA
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 16]; Test type: Superiority or Other; p = 0.9386, ANOVA
Statistical Analysis 19: Comparison: Pregabalin 50 mg vs Placebo; Day 4 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.4352, ANOVA
Statistical Analysis 20: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; p = 0.4522, ANOVA
Statistical Analysis 21: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; p = 0.6606, ANOVA
Statistical Analysis 22: Comparison: Pregabalin 50 mg vs Placebo; Day 5 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.1733, ANOVA
Statistical Analysis 23: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; p = 0.8788, ANOVA
Statistical Analysis 24: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; p = 0.8474, ANOVA
Statistical Analysis 25: Comparison: Pregabalin 50 mg vs Placebo; Day 6 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2938, ANOVA
Statistical Analysis 26: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; p = 0.7602, ANOVA
Statistical Analysis 27: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; p = 0.6881, ANOVA
Statistical Analysis 28: Comparison: Pregabalin 50 mg vs Placebo; Day 7 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.7883, ANOVA
Statistical Analysis 29: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 28]; Test type: Superiority or Other; p = 0.5374, ANOVA
Statistical Analysis 30: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 28]; Test type: Superiority or Other; p = 0.9774, ANOVA
Statistical Analysis 31: Comparison: Pregabalin 50 mg vs Placebo; Day 8 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.3082, ANOVA
Statistical Analysis 32: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 31]; Test type: Superiority or Other; p = 0.4373, ANOVA
Statistical Analysis 33: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 31]; Test type: Superiority or Other; p = 0.6540, ANOVA
Statistical Analysis 34: Comparison: Pregabalin 50 mg vs Placebo; Day 9 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0002, ANOVA
Statistical Analysis 35: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 34]; Test type: Superiority or Other; p = 0.0696, ANOVA
Statistical Analysis 36: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 34]; Test type: Superiority or Other; p = 0.0029, ANOVA
Statistical Analysis 37: Comparison: Pregabalin 50 mg vs Placebo; Day 10 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.3695, ANOVA
Statistical Analysis 38: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 37]; Test type: Superiority or Other; p = 0.9346, ANOVA
Statistical Analysis 39: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 37]; Test type: Superiority or Other; p = 0.9631, ANOVA

7. Secondary Outcome: Numeric Rating Scale (NRS): Current Pain at Rest - Area Under the Curve (AUC)
Description: NRS: a self-administered questionnaire to rate pain. AUC for a single item asking participant to rate current pain at rest (preceding pain with movement); range: 0 (no pain) to 10 (worst pain).
Time Frame: 1 through 48 hours post surgery (PS)
Population: MITT; data from 1 site excluded due to GCP deviations.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
score on scale | 133.8 (7.88) | 141.3 (7.99) | 132.3 (7.78) | 135.1 (7.86)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers. Last observation carried forward or first non-missing observation carried backward algorithm applied to missing scores 1-3 h PS and independently to missing scores 24-48 h PS, before applying trapezoidal rule to compute AUC. AUC=missing if all scores 1-3 or 24-48 h PS missing; Test type: Superiority or Other; p = 0.9025, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.5652, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.7920, ANOVA

8. Secondary Outcome: Numeric Rating Scale (NRS): Average Pain
Description: NRS: a self-administered questionnaire to rate pain. A single item asks participant to rate pain on average in the last 24 hours; range: 0 (no pain) to 10 (worst pain).
Time Frame: 2 hours (h) before surgery (BS); 1, 2, and 3 h post surgery (PS); Days 1, 2, 3, 4, 5, 6, and 7 PS
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on scale
  2 h BS (n=102, 99, 101, 101) | 1.3 (0.15) | 1.3 (0.15) | 1.3 (0.15) | 1.4 (0.15)
  1 h PS (n=101, 96, 99, 99) | 2.8 (0.19) | 3.0 (0.20) | 2.5 (0.19) | 3.2 (0.19)
  2 h PS (n=101, 97, 101, 99) | 3.0 (0.18) | 3.2 (0.18) | 2.8 (0.18) | 3.1 (0.18)
  3 h PS (n=102, 99, 101, 101) | 2.8 (0.17) | 3.2 (0.18) | 2.9 (0.17) | 3.2 (0.17)
  Day 1 PS (n=101, 99, 101, 99) | 3.4 (0.20) | 3.4 (0.20) | 2.9 (0.20) | 3.4 (0.20)
  Day 2 PS (n=102, 99, 99, 100) | 2.9 (0.19) | 3.1 (0.19) | 2.9 (0.19) | 2.9 (0.19)
  Day 3 PS (n=102, 98, 98 101) | 2.5 (0.18) | 2.5 (0.18) | 2.4 (0.18) | 2.5 (0.18)
  Day 4 PS (n=101, 99, 97, 100) | 1.9 (0.17) | 2.0 (0.17) | 2.1 (0.17) | 1.9 (0.17)
  Day 5 PS (n=101, 99, 98, 100) | 1.6 (0.15) | 1.8 (0.15) | 1.7 (0.15) | 1.8 (0.15)
  Day 6 PS (n=98, 96, 91, 96) | 1.4 (0.14) | 1.5 (0.14) | 1.7 (0.14) | 1.6 (0.14)
  Day 7 PS (n=63, 66, 56, 62) | 1.6 (0.19) | 1.5 (0.18) | 1.4 (0.20) | 1.3 (0.19)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.6679, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.7308, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.6781, ANOVA
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.0930, ANOVA
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.3751, ANOVA
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.0111, ANOVA
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.6811, ANOVA
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.7426, ANOVA
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.1619, ANOVA
Statistical Analysis 10: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.1132, ANOVA
Statistical Analysis 11: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.9822, ANOVA
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.1883, ANOVA
Statistical Analysis 13: Comparison: Pregabalin 50 mg vs Placebo; Day 1 PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.9391, ANOVA
Statistical Analysis 14: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.9664, ANOVA
Statistical Analysis 15: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.0747, ANOVA
Statistical Analysis 16: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.9681, ANOVA
Statistical Analysis 17: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.3246, ANOVA
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.7984, ANOVA
Statistical Analysis 19: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 6, analysis 16]; Test type: Superiority or Other; p = 0.8581, ANOVA
Statistical Analysis 20: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 16]; Test type: Superiority or Other; p = 0.9677, ANOVA
Statistical Analysis 21: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 16]; Test type: Superiority or Other; p = 0.7104, ANOVA
Statistical Analysis 22: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; p = 0.8978, ANOVA
Statistical Analysis 23: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; p = 0.6260, ANOVA
Statistical Analysis 24: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; p = 0.4047, ANOVA
Statistical Analysis 25: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; p = 0.4461, ANOVA
Statistical Analysis 26: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; p = 0.9099, ANOVA
Statistical Analysis 27: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; p = 0.8805, ANOVA
Statistical Analysis 28: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; p = 0.2348, ANOVA
Statistical Analysis 29: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; p = 0.4445, ANOVA
Statistical Analysis 30: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; p = 0.8849, ANOVA
Statistical Analysis 31: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 6, analysis 28]; Test type: Superiority or Other; p = 0.2796, ANOVA
Statistical Analysis 32: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 6, analysis 28]; Test type: Superiority or Other; p = 0.5225, ANOVA
Statistical Analysis 33: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 6, analysis 28]; Test type: Superiority or Other; p = 0.7015, ANOVA

9. Secondary Outcome: Time From End of Surgery to First Rescue Medication
Description: Rescue medication includes both naproxen and narcotic medication (including tramadol and opioid analgesics). For subjects without use of rescue medication, the time-to-event variable is censored at the Beginning of Taper Visit (Day 7 PS) or at time of withdrawal.
Time Frame: Day 1 through Day 7 post surgery
Population: MITT; data from 1 site excluded due to GCP deviations. No descriptive statistics were generated.
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Time From End of Surgery to Reach a Total Score of at Least 9 on the Post-Anesthetic Discharge Scoring System (PADS)
Description: PADS is a 5-item scale (individual item range: 0-2; higher scores indicating better readiness for hospital discharge). Total score range: 0-10, with 9 or higher indicating eligibility for discharge. End of surgery is time of transfer to post-anesthesia care unit (PACU). Subjects who did not reach a score of 9 on PADS were censored at the date and time of discharge.
Time Frame: Day 1
Population: MITT; data from 1 site excluded due to GCP deviations. No descriptive statistics were generated.
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Time From End of Surgery to Discharge From Post-Anesthesia Care Unit (PACU)
Time Frame: Day 1
Population: MITT; data from 1 site excluded due to GCP deviations. Data not analyzed as planned.
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Daily Sleep Interference Rating Scale (DSIRS) Score
Description: DSIRS: self-administered 11-point Likert scale ranging from 0 (pain does not interfere with sleep) to 10 (pain completely interferes with sleep [unable to sleep due to pain]) during past 24-hour period. Higher score indicates a greater level of sleep disturbance. Performed daily on awakening, prior to taking study medication.
Time Frame: Days 2, 3, 4, 5, 6, 7, 8, 9, and 10 post surgery (PS)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on a scale
  Day 2 PS (n=102, 99, 101, 101) | 2.86 (0.250) | 2.61 (0.255) | 2.17 (0.250) | 3.18 (0.251)
  Day 3 PS (n=102, 98, 100, 101) | 2.13 (0.211) | 2.01 (0.216) | 1.50 (0.213) | 2.11 (0.212)
  Day 4 PS (n=101, 99, 99, 101) | 1.52 (0.199) | 1.40 (0.201) | 1.27 (0.200) | 1.48 (0.198)
  Day 5 PS (n=101, 98, 98, 100) | 1.03 (0.172) | 1.22 (0.174) | 1.09 (0.173) | 1.44 (0.172)
  Day 6 PS (n=100, 99, 98, 99) | 0.94 (0.147) | 0.98 (0.147) | 0.81 (0.147) | 1.13 (0.147)
  Day 7 PS (n=98, 96, 92, 96) | 1.04 (0.150) | 0.90 (0.151) | 0.72 (0.154) | 1.00 (0.150)
  Day 8 PS (n=61, 65, 54, 61) | 1.00 (0.185) | 0.90 (0.180) | 0.59 (0.202) | 0.63 (0.185)
  Day 9 PS (n=21, 24, 25, 24) | 0.14 (0.240) | 1.01 (0.222) | 0.40 (0.222) | 1.01 (0.212)
  Day 10 PS (n=11, 11, 13, 11) | 0.15 (0.349) | 1.16 (0.347) | 0.08 (0.332) | 0.72 (0.310)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; Day 2 PS; LS Means from ANOVA model with terms of treatment, pooled center. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.3332, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.0933, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.0031, ANOVA
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; Day 3 PS; LS Means from ANOVA model with terms of treatment, pooled center. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.9451, ANOVA
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 12, analysis 4]; Test type: Superiority or Other; p = 0.7312, ANOVA
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 12, analysis 4]; Test type: Superiority or Other; p = 0.0348, ANOVA
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; Day 4 PS; LS Means from ANOVA model with terms of treatment, pooled center. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.8936, ANOVA
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p = 0.7672, ANOVA
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p = 0.4285, ANOVA
Statistical Analysis 10: Comparison: Pregabalin 50 mg vs Placebo; Day 5 PS; LS Means from ANOVA model with terms of treatment, pooled center. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0785, ANOVA
Statistical Analysis 11: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 12, analysis 10]; Test type: Superiority or Other; p = 0.3348, ANOVA
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 12, analysis 10]; Test type: Superiority or Other; p = 0.1366, ANOVA
Statistical Analysis 13: Comparison: Pregabalin 50 mg vs Placebo; Day 6 PS; LS Means from ANOVA model with terms of treatment, pooled center. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.3338, ANOVA
Statistical Analysis 14: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 12, analysis 13]; Test type: Superiority or Other; p = 0.4460, ANOVA
Statistical Analysis 15: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 12, analysis 13]; Test type: Superiority or Other; p = 0.1078, ANOVA
Statistical Analysis 16: Comparison: Pregabalin 50 mg vs Placebo; Day 7 PS; LS Means from ANOVA model with terms of treatment, pooled center. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.8273, ANOVA
Statistical Analysis 17: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 12, analysis 16]; Test type: Superiority or Other; p = 0.6140, ANOVA
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 12, analysis 16]; Test type: Superiority or Other; p = 0.1684, ANOVA
Statistical Analysis 19: Comparison: Pregabalin 50 mg vs Placebo; Day 8 PS; LS Means from ANOVA model with terms of treatment, pooled center. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.1285, ANOVA
Statistical Analysis 20: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 12, analysis 19]; Test type: Superiority or Other; p = 0.2640, ANOVA
Statistical Analysis 21: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 12, analysis 19]; Test type: Superiority or Other; p = 0.8956, ANOVA
Statistical Analysis 22: Comparison: Pregabalin 50 mg vs Placebo; Day 9 PS; LS Means from ANOVA model with terms of treatment, pooled center. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0058, ANOVA
Statistical Analysis 23: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 12, analysis 22]; Test type: Superiority or Other; p = 0.9929, ANOVA
Statistical Analysis 24: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 12, analysis 22]; Test type: Superiority or Other; p = 0.0473, ANOVA
Statistical Analysis 25: Comparison: Pregabalin 50 mg vs Placebo; Day 10 PS; LS Means from ANOVA model with terms of treatment, pooled center. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2426, ANOVA
Statistical Analysis 26: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 12, analysis 25]; Test type: Superiority or Other; p = 0.3478, ANOVA
Statistical Analysis 27: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 12, analysis 25]; Test type: Superiority or Other; p = 0.1694, ANOVA

13. Secondary Outcome: Total Cumulative Dose of Opioids and Tramadol Used During and After Surgery
Description: Total cumulative dose of opioids and tramadol administered by any route during surgery and postoperatively. Dose of tramadol calculated as milligrams (mg) of oral morphine equivalent.
Time Frame: 24, 48, and 72 hours (h) post surgery (PS), and Days 4, 5, 6, and 7 PS
Population: MITT; data from 1 site excluded due to GCP deviations; n=number of subjects with analyzable data at observation (pregabalin 50 mg, pregabalin 150 mg, pregabalin 300 mg, and placebo, respectively). During surgery data not analyzed as planned.
Measure: Least Squares Mean (Standard Error); unit: mg
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
mg
  24 h PS (n=102, 99, 101, 101) | 10.29 (2.275) | 9.44 (2.320) | 6.58 (2.279) | 16.03 (2.283)
  48 h PS (n=102, 99, 101, 101) | 13.15 (2.763) | 14.10 (2.817) | 9.73 (2.768) | 19.79 (2.772)
  72 h PS (n=102, 99, 101, 101) | 14.59 (3.088) | 16.99 (3.148) | 12.34 (3.092) | 22.20 (3.097)
  Day 4 PS (n=102, 99, 101, 101) | 15.35 (3.474) | 18.65 (3.542) | 14.18 (3.479) | 23.97 (3.485)
  Day 5 PS (n=102, 99, 101, 101) | 16.09 (3.786) | 20.46 (3.860) | 14.64 (3.792) | 25.57 (3.798)
  Day 6 PS (n=101, 99, 99, 100) | 15.99 (4.072) | 21.57 (4.139) | 15.81 (4.105) | 26.90 (4.085)
  Day 7 PS (n=99, 99, 97, 100) | 15.88 (4.291) | 22.23 (4.322) | 16.16 (4.334) | 28.15 (4.265)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; 24 h PS; LS Means from ANOVA model with terms of treatment, pooled center. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0630, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0347, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0024, ANOVA
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; 48 h PS; LS Means from ANOVA model with terms of treatment, pooled center. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0767, ANOVA
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 13, analysis 4]; Test type: Superiority or Other; p = 0.1327, ANOVA
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 13, analysis 4]; Test type: Superiority or Other; p = 0.0078, ANOVA
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; 72 h PS; LS Means from ANOVA model with terms of treatment, pooled center. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0694, ANOVA
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p = 0.2173, ANOVA
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p = 0.0193, ANOVA
Statistical Analysis 10: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p = 0.0673, ANOVA
Statistical Analysis 11: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p = 0.2629, ANOVA
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p = 0.0388, ANOVA
Statistical Analysis 13: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 12, analysis 10]; Test type: Superiority or Other; p = 0.0651, ANOVA
Statistical Analysis 14: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 12, analysis 10]; Test type: Superiority or Other; p = 0.3242, ANOVA
Statistical Analysis 15: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 12, analysis 10]; Test type: Superiority or Other; p = 0.0345, ANOVA
Statistical Analysis 16: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 12, analysis 13]; Test type: Superiority or Other; p = 0.0487, ANOVA
Statistical Analysis 17: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 12, analysis 13]; Test type: Superiority or Other; p = 0.3384, ANOVA
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 12, analysis 13]; Test type: Superiority or Other; p = 0.0467, ANOVA
Statistical Analysis 19: Comparison: Pregabalin 50 mg vs Placebo; [analysis description as in outcome 12, analysis 16]; Test type: Superiority or Other; p = 0.0347, ANOVA
Statistical Analysis 20: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 12, analysis 16]; Test type: Superiority or Other; p = 0.3086, ANOVA
Statistical Analysis 21: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 12, analysis 16]; Test type: Superiority or Other; p = 0.0406, ANOVA

14. Secondary Outcome: Amount of Non-opioid Rescue Medication (Naproxen and Antiemetic Medications) Used During the Study
Description: Total cumulative dose of naproxen calculated in milligrams (mg) from the end of surgery up to and including Day 7 after surgery.
Time Frame: End of Surgery through Day 7 post surgery
Population: MITT; data from 1 site excluded due to GCP deviations. Amount of antiemetic rescue medications not analyzed as planned.
Measure: Least Squares Mean (Standard Error); unit: mg
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
mg | 3938.81 (155.124) | 3930.57 (155.304) | 3892.96 (154.413) | 3770.07 (153.322)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.4177, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.4410, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.5560, ANOVA

15. Secondary Outcome: Total Clinically Meaningful Event (CME) Score and Cumulative Total Distinct CME Score Using the Opioid-Related Symptom Distress Scale (OR-SDS)
Description: OR-SDS: a self-administered assessment of 10 common opioid-related side effects (symptoms). A CME is a severe or very severe symptom (or moderate or greater severity symptom of confusion). The Total Distinct CME score is the sum of CMEs across symptoms (range: 0 [none] to 10 [10 CMEs]); the Cumulative Total Distinct (CT Distinct) CME score is the sum of Total Distinct CME scores at observation and prior observations. The Total CME score is the same as the Total Distinct CME score except that only 1 CME is counted if both nausea and vomiting (or retching) occur (range: 0 [none] to 9 [9 CMEs]).
Time Frame: 3, 24, and 72 hours (h) Post-Surgery (PS), and End of Treatment (EOT [Day 7 PS or Early Termination])
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on a scale
  Total CME 3 h PS (n=98, 97, 98, 98) | 0.2 (0.07) | 0.2 (0.07) | 0.1 (0.07) | 0.2 (0.07)
  Total CME 24 h PS (n=97, 97, 98, 97) | 0.2 (0.07) | 0.3 (0.07) | 0.4 (0.07) | 0.2 (0.07)
  Total CME 72 h PS (n=98, 96, 96, 96) | 0.1 (0.05) | 0.1 (0.05) | 0.2 (0.05) | 0.1 (0.05)
  Total CME EOT (n=100, 98, 99, 97) | 0.0 (0.04) | 0.1 (0.04) | 0.1 (0.04) | 0.1 (0.04)
  CT Distinct CME 3 h PS (n=98, 97, 98, 98) | 0.2 (0.07) | 0.2 (0.07) | 0.1 (0.07) | 0.2 (0.07)
  CT Distinct CME 24 h PS (n=93, 95, 96, 94) | 0.3 (0.10) | 0.4 (0.10) | 0.4 (0.09) | 0.4 (0.10)
  CT Distinct CME 72 h PS (n=91, 92, 93, 92) | 0.3 (0.11) | 0.5 (0.11) | 0.5 (0.11) | 0.5 (0.11)
  CT Distinct CME EOT (n=90, 92, 93, 89) | 0.3 (0.11) | 0.5 (0.11) | 0.6 (0.11) | 0.6 (0.11)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; Total CME 3 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.4273, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.4466, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.3785, ANOVA
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; Total CME 24 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.5272, ANOVA
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 15, analysis 4]; Test type: Superiority or Other; p = 0.4257, ANOVA
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 15, analysis 4]; Test type: Superiority or Other; p = 0.1428, ANOVA
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; Total CME 72 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2316, ANOVA
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 15, analysis 7]; Test type: Superiority or Other; p = 0.3468, ANOVA
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 15, analysis 7]; Test type: Superiority or Other; p = 0.5367, ANOVA
Statistical Analysis 10: Comparison: Pregabalin 50 mg vs Placebo; Total CME EOT; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0549, ANOVA
Statistical Analysis 11: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 15, analysis 10]; Test type: Superiority or Other; p = 0.1351, ANOVA
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 15, analysis 10]; Test type: Superiority or Other; p = 0.9599, ANOVA
Statistical Analysis 13: Comparison: Pregabalin 50 mg vs Placebo; CT Distinct CME 3 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.4273, ANOVA
Statistical Analysis 14: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.4466, ANOVA
Statistical Analysis 15: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.3785, ANOVA
Statistical Analysis 16: Comparison: Pregabalin 50 mg vs Placebo; CT Distinct CME 24 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2869, ANOVA
Statistical Analysis 17: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 15, analysis 16]; Test type: Superiority or Other; p = 0.9905, ANOVA
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 15, analysis 16]; Test type: Superiority or Other; p = 0.9381, ANOVA
Statistical Analysis 19: Comparison: Pregabalin 50 mg vs Placebo; CT Distinct CME 72 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2158, ANOVA
Statistical Analysis 20: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 15, analysis 19]; Test type: Superiority or Other; p = 0.7887, ANOVA
Statistical Analysis 21: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 15, analysis 19]; Test type: Superiority or Other; p = 0.9250, ANOVA
Statistical Analysis 22: Comparison: Pregabalin 50 mg vs Placebo; CT Distinct CME EOT; LS Means from ANOVA model with terms of treatment, pooled center and baseline pain catastrophizing total score. Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.1472, ANOVA
Statistical Analysis 23: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 15, analysis 22]; Test type: Superiority or Other; p = 0.5383, ANOVA
Statistical Analysis 24: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 15, analysis 22]; Test type: Superiority or Other; p = 0.8869, ANOVA

16. Secondary Outcome: Participants With Clinically Meaningful Events (CMEs) for Individual Symptoms Using the Opioid-Related Symptom Distress Scale (OR-SDS)
Description: OR-SDS: a self-administered assessment of 10 common opioid-related side effects (symptoms). A CME is a severe or very severe symptom (or moderate or greater severity symptom of confusion). For individual symptom categories, the number of subjects who experienced at least one CME. Concentrate (concentr).
Time Frame: 3, 24, and 72 hours (h) post surgery (PS), and End of Treatment (EOT [Day 7 PS or Early Termination])
Population: MITT; data from 1 site excluded due to GCP deviations.
Measure: Number; unit: participants
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
participants
  Fatigue 3 h PS (n=99, 98, 98, 100) | 4 | 2 | 2 | 2
  Fatigue 24 h PS (n=99, 97, 100, 97) | 2 | 3 | 6 | 2
  Fatigue 72 h PS (n=101, 97, 98, 98) | 0 | 0 | 1 | 1
  Fatigue EOT (n=100, 98, 100, 98) | 0 | 0 | 0 | 3
  Drowsiness 3 h PS (n=99, 98, 98, 100) | 5 | 4 | 4 | 4
  Drowsiness 24 h PS (n=98, 98, 99, 97) | 2 | 7 | 8 | 3
  Drowsiness 72 h PS (n=100, 98, 98, 98) | 1 | 0 | 1 | 3
  Drowsiness EOT (n=100, 98, 100, 97) | 0 | 0 | 2 | 3
  Inability to concentr 3 h PS (n=100, 97, 98, 99) | 1 | 0 | 0 | 2
  Inability to concentr 24 h PS (n=99, 98, 100, 97) | 1 | 1 | 2 | 2
  Inability to concentr 72 h PS (101, 98, 98, 97) | 0 | 0 | 1 | 1
  Inability to concentr EOT (n=100, 98, 100, 99) | 1 | 0 | 0 | 1
  Nausea 3 h PS (n=101, 97, 99, 100) | 2 | 1 | 1 | 4
  Nausea 24 h PS (n=100, 99, 101, 98) | 3 | 4 | 3 | 1
  Nausea 72 h PS (n=101, 99, 99, 98) | 0 | 0 | 0 | 0
  Nausea EOT (n=101, 98, 100, 99) | 1 | 0 | 2 | 1
  Dizziness 3 h PS (n=101, 97, 99, 100) | 2 | 1 | 5 | 6
  Dizziness 24 h PS (n=100, 98, 99, 98) | 2 | 3 | 6 | 1
  Dizziness 72 h PS (n=101, 98, 97, 98) | 0 | 0 | 1 | 0
  Dizziness EOT (n=101, 98, 100, 99) | 1 | 0 | 1 | 0
  Constipation 3 h PS (n=101, 98, 99, 100) | 1 | 0 | 0 | 1
  Constipation 24 h PS (n=99, 99, 100, 98) | 4 | 4 | 7 | 5
  Constipation 72 h PS (n=99, 97, 98, 98) | 4 | 7 | 10 | 7
  Constipation EOT (n=101, 98, 99, 99) | 1 | 2 | 5 | 2
  Itching 3 h PS (n=100, 98, 99, 100) | 0 | 1 | 0 | 0
  Itching 24 h PS (n=100, 99, 101, 98) | 0 | 0 | 1 | 1
  Itching 72 h PS (n=100, 99, 99, 97) | 1 | 1 | 0 | 1
  Itching EOT (n=101, 98, 100, 98) | 0 | 0 | 0 | 1
  Difficulty Urinating 3 h PS (n=101, 98, 99, 99) | 0 | 3 | 2 | 1
  Difficulty Urinating 24 h PS (n=100, 99, 100, 98) | 2 | 4 | 5 | 3
  Difficulty Urinating 72 h PS (n=100, 99, 99, 98) | 2 | 0 | 3 | 0
  Difficulty Urinating EOT (n= 101, 98, 100, 99) | 1 | 0 | 3 | 0
  Confusion 3 h PS (n=101, 98, 99, 100) | 2 | 3 | 3 | 2
  Confusion 24 h PS (n=101, 99, 99, 98) | 1 | 1 | 2 | 1
  Confusion 72 h PS (n=100, 99, 99, 98) | 2 | 1 | 3 | 2
  Confusion EOT (n=101, 98, 100, 99) | 0 | 2 | 0 | 2
  Retching/Vomiting 3 h PS (n=101, 98, 99, 100) | 0 | 0 | 0 | 3
  Retching/Vomiting 24 h PS (n=101, 99, 100, 98) | 0 | 2 | 0 | 1
  Retching/Vomiting 72 h PS (n=101, 99, 99, 98) | 0 | 0 | 0 | 0
  Retching/Vomiting EOT (n=101, 98, 100, 99) | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; Fatigue at 3 h PS;; Test type: Superiority or Other; p = 0.4024, Cochran-Mantel-Haenszel — P-values are derived from CMH test adjusted for pooled centers. Centers with fewer than 8 treated subjects were combined into pooled centers
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; Fatigue at 3 h PS;; Test type: Superiority or Other; p = 0.9766, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; Fatigue at 3 h PS;; Test type: Superiority or Other; p = 0.9975, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; Fatigue at 24 h PS;; Test type: Superiority or Other; p = 0.9038, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; Fatigue at 24 h PS;; Test type: Superiority or Other; p = 0.9370, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; Fatigue at 24 h PS;; Test type: Superiority or Other; p = 0.2134, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; Fatigue at 72 h PS;; Test type: Superiority or Other; p = 0.2482, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; Fatigue at 72 h PS;; Test type: Superiority or Other; p = 0.2207, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; Fatigue at 72 h PS;; Test type: Superiority or Other; p = 0.9191, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 10: Comparison: Pregabalin 50 mg vs Placebo; Fatigue at EOT;; Test type: Superiority or Other; p = 0.0686, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 11: Comparison: Pregabalin 150 mg vs Placebo; Fatigue at EOT;; Test type: Superiority or Other; p = 0.0746, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; Fatigue at EOT;; Test type: Superiority or Other; p = 0.0512, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 13: Comparison: Pregabalin 50 mg vs Placebo; Drowsiness at 3 h PS;; Test type: Superiority or Other; p = 0.7118, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 14: Comparison: Pregabalin 150 mg vs Placebo; Drowsiness at 3 h PS;; Test type: Superiority or Other; p = 0.9883, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 15: Comparison: Pregabalin 300 mg vs Placebo; Drowsiness at 3 h PS;; Test type: Superiority or Other; p = 0.9770, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 16: Comparison: Pregabalin 50 mg vs Placebo; Drowsiness at 24 h PS;; Test type: Superiority or Other; p = 0.5457, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 17: Comparison: Pregabalin 150 mg vs Placebo; Drowsiness at 24 h PS;; Test type: Superiority or Other; p = 0.2579, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; Drowsiness at 24 h PS;; Test type: Superiority or Other; p = 0.1232, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 19: Comparison: Pregabalin 50 mg vs Placebo; Drowsiness at 72 h PS;; Test type: Superiority or Other; p = 0.2880, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 20: Comparison: Pregabalin 150 mg vs Placebo; Drowsiness at 72 h PS;; Test type: Superiority or Other; p = 0.0894, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 21: Comparison: Pregabalin 300 mg vs Placebo; Drowsiness at 72 h PS;; Test type: Superiority or Other; p = 0.1979, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 22: Comparison: Pregabalin 50 mg vs Placebo; Drowsiness at EOT;; Test type: Superiority or Other; p = 0.0686, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 23: Comparison: Pregabalin 150 mg vs Placebo; Drowsiness at EOT;; Test type: Superiority or Other; p = 0.0746, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 24: Comparison: Pregabalin 300 mg vs Placebo; Drowsiness at EOT;; Test type: Superiority or Other; p = 0.4669, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 25: Comparison: Pregabalin 50 mg vs Placebo; Inability to Concentrate at 3 h PS;; Test type: Superiority or Other; p = 0.5533, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 26: Comparison: Pregabalin 150 mg vs Placebo; Inability to Concentrate at 3 h PS;; Test type: Superiority or Other; p = 0.1611, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 27: Comparison: Pregabalin 300 mg vs Placebo; Inability to Concentrate at 3 h PS;; Test type: Superiority or Other; p = 0.1611, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 28: Comparison: Pregabalin 50 mg vs Placebo; Inability to Concentrate at 24 h PS;; Test type: Superiority or Other; p = 0.4793, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 29: Comparison: Pregabalin 150 mg vs Placebo; Inability to Concentrate at 24 h PS;; Test type: Superiority or Other; p = 0.3533, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 30: Comparison: Pregabalin 300 mg vs Placebo; Inability to Concentrate at 24 h PS;; Test type: Superiority or Other; p = 0.8852, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 31: Comparison: Pregabalin 50 mg vs Placebo; Inability to Concentrate at 72 h PS;; Test type: Superiority or Other; p = 0.3173, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 32: Comparison: Pregabalin 150 mg vs Placebo; Inability to Concentrate at 72 h PS;; Test type: Superiority or Other; p = 0.3173, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 33: Comparison: Pregabalin 300 mg vs Placebo; Inability to Concentrate at 72 h PS;; Test type: Superiority or Other; p = 0.8864, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 34: Comparison: Pregabalin 50 mg vs Placebo; Inability to Concentrate at EOT;; Test type: Superiority or Other; p = 0.8084, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 35: Comparison: Pregabalin 150 mg vs Placebo; Inability to Concentrate at EOT;; Test type: Superiority or Other; p = 0.3173, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 36: Comparison: Pregabalin 300 mg vs Placebo; Inability to Concentrate at EOT;; Test type: Superiority or Other; p = 0.2207, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 37: Comparison: Pregabalin 50 mg vs Placebo; Nausea at 3 h PS;; Test type: Superiority or Other; p = 0.3747, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 38: Comparison: Pregabalin 150 mg vs Placebo; Nausea at 3 h PS;; Test type: Superiority or Other; p = 0.1450, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 39: Comparison: Pregabalin 300 mg vs Placebo; Nausea at 3 h PS;; Test type: Superiority or Other; p = 0.2054, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 40: Comparison: Pregabalin 50 mg vs Placebo; Nausea at 24 h PS;; Test type: Superiority or Other; p = 0.4106, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 41: Comparison: Pregabalin 150 mg vs Placebo; Nausea at 24 h PS;; Test type: Superiority or Other; p = 0.2199, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 42: Comparison: Pregabalin 300 mg vs Placebo; Nausea at 24 h PS;; Test type: Superiority or Other; p = 0.2896, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 43: Comparison: Pregabalin 50 mg vs Placebo; Nausea at EOT;; Test type: Superiority or Other; p = 1.0000, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 44: Comparison: Pregabalin 150 mg vs Placebo; Nausea at EOT;; Test type: Superiority or Other; p = 0.3173, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 45: Comparison: Pregabalin 300 mg vs Placebo; Nausea at EOT;; Test type: Superiority or Other; p = 0.3943, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 46: Comparison: Pregabalin 50 mg vs Placebo; Dizziness at 3 h PS;; Test type: Superiority or Other; p = 0.1703, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 47: Comparison: Pregabalin 150 mg vs Placebo; Dizziness at 3 h PS;; Test type: Superiority or Other; p = 0.0807, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 48: Comparison: Pregabalin 300 mg vs Placebo; Dizziness at 3 h PS;; Test type: Superiority or Other; p = 0.7728, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 49: Comparison: Pregabalin 50 mg vs Placebo; Dizziness at 24 h PS;; Test type: Superiority or Other; p = 0.4770, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 50: Comparison: Pregabalin 150 mg vs Placebo; Dizziness at 24 h PS;; Test type: Superiority or Other; p = 0.3625, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 51: Comparison: Pregabalin 300 mg vs Placebo; Dizziness at 24 h PS;; Test type: Superiority or Other; p = 0.0617, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 52: Comparison: Pregabalin 300 mg vs Placebo; Dizziness at 72 h PS;; Test type: Superiority or Other; p = 0.3061, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 53: Comparison: Pregabalin 50 mg vs Placebo; Dizziness at EOT;; Test type: Superiority or Other; p = 0.2207, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 54: Comparison: Pregabalin 300 mg vs Placebo; Dizziness at EOT;; Test type: Superiority or Other; p = 0.3173, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 55: Comparison: Pregabalin 50 mg vs Placebo; Constipation at 3 h PS;; Test type: Superiority or Other; p = 0.9191, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 56: Comparison: Pregabalin 150 mg vs Placebo; Constipation at 3 h PS;; Test type: Superiority or Other; p = 0.3173, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 57: Comparison: Pregabalin 300 mg vs Placebo; Constipation at 3 h PS;; Test type: Superiority or Other; p = 0.2207, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 58: Comparison: Pregabalin 50 mg vs Placebo; Constipation at 24 h PS;; Test type: Superiority or Other; p = 0.6692, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 59: Comparison: Pregabalin 150 mg vs Placebo; Constipation at 24 h PS;; Test type: Superiority or Other; p = 0.7793, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 60: Comparison: Pregabalin 300 mg vs Placebo; Constipation at 24 h PS;; Test type: Superiority or Other; p = 0.6065, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 61: Comparison: Pregabalin 50 mg vs Placebo; Constipation at 72 h PS;; Test type: Superiority or Other; p = 0.3570, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 62: Comparison: Pregabalin 150 mg vs Placebo; Constipation at 72 h PS;; Test type: Superiority or Other; p = 0.9690, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 63: Comparison: Pregabalin 300 mg vs Placebo; Constipation at 72 h PS;; Test type: Superiority or Other; p = 0.5299, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 64: Comparison: Pregabalin 50 mg vs Placebo; Constipation at EOT;; Test type: Superiority or Other; p = 0.4821, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 65: Comparison: Pregabalin 150 mg vs Placebo; Constipation at EOT;; Test type: Superiority or Other; p = 0.8295, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 66: Comparison: Pregabalin 300 mg vs Placebo; Constipation at EOT;; Test type: Superiority or Other; p = 0.3304, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 67: Comparison: Pregabalin 150 mg vs Placebo; Itching at 3 h PS;; Test type: Superiority or Other; p = 0.2482, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 68: Comparison: Pregabalin 50 mg vs Placebo; Itching at 24 h PS;; Test type: Superiority or Other; p = 0.2482, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 69: Comparison: Pregabalin 150 mg vs Placebo; Itching at 24 h PS;; Test type: Superiority or Other; p = 0.2207, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 70: Comparison: Pregabalin 300 mg vs Placebo; Itching at 24 h PS;; Test type: Superiority or Other; p = 0.8055, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 71: Comparison: Pregabalin 50 mg vs Placebo; Itching at 72 h PS;; Test type: Superiority or Other; p = 0.9191, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 72: Comparison: Pregabalin 150 mg vs Placebo; Itching at 72 h PS;; Test type: Superiority or Other; p = 0.8488, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 73: Comparison: Pregabalin 300 mg vs Placebo; Itching at 72 h PS;; Test type: Superiority or Other; p = 0.2482, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 74: Comparison: Pregabalin 50 mg vs Placebo; Itching at EOT;; Test type: Superiority or Other; p = 0.2482, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 75: Comparison: Pregabalin 150 mg vs Placebo; Itching at EOT;; Test type: Superiority or Other; p = 0.2207, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 76: Comparison: Pregabalin 300 mg vs Placebo; Itching at EOT;; Test type: Superiority or Other; p = 0.2482, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 77: Comparison: Pregabalin 50 mg vs Placebo; Difficulty Urinating at 3 h PS;; Test type: Superiority or Other; p = 0.3291, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 78: Comparison: Pregabalin 150 mg vs Placebo; Difficulty Urinating at 3 h PS;; Test type: Superiority or Other; p = 0.1391, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 79: Comparison: Pregabalin 300 mg vs Placebo; Difficulty Urinating at 3 h PS;; Test type: Superiority or Other; p = 0.6318, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 80: Comparison: Pregabalin 50 mg vs Placebo; Difficulty Urinating at 24 h PS;; Test type: Superiority or Other; p = 0.6319, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 81: Comparison: Pregabalin 150 mg vs Placebo; Difficulty Urinating at 24 h PS;; Test type: Superiority or Other; p = 0.8149, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 82: Comparison: Pregabalin 300 mg vs Placebo; Difficulty Urinating at 24 h PS;; Test type: Superiority or Other; p = 0.5795, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 83: Comparison: Pregabalin 50 mg vs Placebo; Difficulty Urinating at 72 h PS;; Test type: Superiority or Other; p = 0.1750, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 84: Comparison: Pregabalin 300 mg vs Placebo; Difficulty Urinating at 72 h PS;; Test type: Superiority or Other; p = 0.0676, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 85: Comparison: Pregabalin 50 mg vs Placebo; Difficulty Urinating at EOT;; Test type: Superiority or Other; p = 0.2943, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 86: Comparison: Pregabalin 300 mg vs Placebo; Difficulty Urinating at EOT;; Test type: Superiority or Other; p = 0.0719, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 87: Comparison: Pregabalin 50 mg vs Placebo; Confusion at 3 h PS;; Test type: Superiority or Other; p = 0.9283, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 88: Comparison: Pregabalin 150 mg vs Placebo; Confusion at 3 h PS;; Test type: Superiority or Other; p = 0.9024, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 89: Comparison: Pregabalin 300 mg vs Placebo; Confusion at 3 h PS;; Test type: Superiority or Other; p = 0.7655, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 90: Comparison: Pregabalin 50 mg vs Placebo; Confusion at 24 h PS;; Test type: Superiority or Other; p = 1.0000, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 91: Comparison: Pregabalin 150 mg vs Placebo; Confusion at 24 h PS;; Test type: Superiority or Other; p = 0.8460, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 92: Comparison: Pregabalin 300 mg vs Placebo; Confusion at 24 h PS;; Test type: Superiority or Other; p = 0.6419, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 93: Comparison: Pregabalin 50 mg vs Placebo; Confusion at 72 h PS;; Test type: Superiority or Other; p = 0.9522, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 94: Comparison: Pregabalin 150 mg vs Placebo; Confusion at 72 h PS;; Test type: Superiority or Other; p = 0.5800, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 95: Comparison: Pregabalin 300 mg vs Placebo; Confusion at 72 h PS;; Test type: Superiority or Other; p = 0.7675, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 96: Comparison: Pregabalin 50 mg vs Placebo; Confusion at EOT;; Test type: Superiority or Other; p = 0.1672, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 97: Comparison: Pregabalin 150 mg vs Placebo; Confusion at EOT;; Test type: Superiority or Other; p = 0.9634, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 98: Comparison: Pregabalin 300 mg vs Placebo; Confusion at EOT;; Test type: Superiority or Other; p = 0.1161, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 99: Comparison: Pregabalin 50 mg vs Placebo; Retching/Vomiting at 3 h PS;; Test type: Superiority or Other; p = 0.0754, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 100: Comparison: Pregabalin 150 mg vs Placebo; Retching/Vomiting at 3 h PS;; Test type: Superiority or Other; p = 0.0711, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 101: Comparison: Pregabalin 300 mg vs Placebo; Retching/Vomiting at 3 h PS;; Test type: Superiority or Other; p = 0.0711, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 102: Comparison: Pregabalin 50 mg vs Placebo; Retching/Vomiting at 24 h PS;; Test type: Superiority or Other; p = 0.2482, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 103: Comparison: Pregabalin 150 mg vs Placebo; Retching/Vomiting at 24 h PS;; Test type: Superiority or Other; p = 0.8091, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 104: Comparison: Pregabalin 300 mg vs Placebo; Retching/Vomiting at 24 h PS;; Test type: Superiority or Other; p = 0.2482, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 105: Comparison: Pregabalin 50 mg vs Placebo; Retching/Vomiting at EOT;; Test type: Superiority or Other; p = 0.3173, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 106: Comparison: Pregabalin 150 mg vs Placebo; Retching/Vomiting at EOT;; Test type: Superiority or Other; p = 0.3173, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 107: Comparison: Pregabalin 300 mg vs Placebo; Retching/Vomiting at EOT;; Test type: Superiority or Other; p = 0.4386, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]

17. Secondary Outcome: Subject Global Evaluation of Study Medication (GESM)
Description: GESM is a self-administered overall impression (global evaluation) of study medication received for pain; 4 categories: poor, fair, good, and excellent.
Time Frame: 24 hours (h) post surgery (PS) and End of Treatment (EOT [Day 7 PS or Early Termination])
Population: MITT; data from 1 site excluded due to GCP deviations
Measure: Number; unit: participants
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
participants
  24 h PS: Poor (n=100, 96, 101, 99) | 10 | 8 | 7 | 15
  24 h PS: Fair (n=100, 96, 101, 99) | 29 | 28 | 25 | 32
  24 h PS: Good (n=100, 96, 101, 99) | 45 | 46 | 42 | 40
  24 h PS: Excellent (n=100, 96, 101, 99) | 16 | 14 | 27 | 12
  EOT: Poor (n=99, 99, 100, 100) | 9 | 10 | 6 | 18
  EOT: Fair (n=99, 99, 100, 100) | 14 | 19 | 14 | 19
  EOT: Good (n=99, 99, 100, 100) | 45 | 37 | 30 | 32
  EOT: Excellent (n=99, 99, 100, 100) | 31 | 33 | 50 | 31
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; 24 h PS; Test type: Superiority or Other; p = 0.1723, Cochran-Mantel-Haenszel — P-values derived from Cochran-Mantel-Haenszel (CMH) test adjusted for pooled centers. Centers with fewer than 8 treated subjects were combined into pooled centers
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; 24 h PS; Test type: Superiority or Other; p = 0.0639, Cochran-Mantel-Haenszel — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; 24 h PS; Test type: Superiority or Other; p = 0.0021, Cochran-Mantel-Haenszel — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; EOT; Test type: Superiority or Other; p = 0.1127, Cochran-Mantel-Haenszel — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; EOT; Test type: Superiority or Other; p = 0.0703, Cochran-Mantel-Haenszel — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; EOT; Test type: Superiority or Other; p = 0.0012, Cochran-Mantel-Haenszel — [p-value comment as in outcome 17, analysis 1]

18. Secondary Outcome: Participants With Wound Healing Complications
Description: Investigator-assigned mutually exclusive categories of: 1) no surgical wound complication, 2) superficial incisional surgical site infection, 3) deep incisional surgical site infection, 4) organ or space surgical site infection, or 5) non-infectious wound healing complication.
Time Frame: Day 7 post surgery (PS) and up to 30 days PS
Population: Operated subjects within the safety population. Safety population=all randomized subjects administered at least 1 dose of study drug and for whom at least 1 post-baseline safety evaluation was obtained.
Measure: Number; unit: participants
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 106 | 104 | 102 | 106
participants
  No surgical wound complication | 102 | 102 | 99 | 101
  Superficial incisional surgical site infection | 1 | 0 | 1 | 1
  Deep incisional surgical site infection | 0 | 0 | 0 | 0
  Organ/space surgical site infection | 0 | 0 | 0 | 0
  Non-infectious wound healing complication | 2 | 1 | 1 | 1

19. Secondary Outcome: Participants With Physician Contacts Post-discharge
Description: Number of participants who answered "yes" to the Post-Surgery Contact question: "From the time you were discharged from the hospital, did you have to contact any type of physician because of pain, difficulty getting up and walking about, or difficulty with passing urine?"
Time Frame: 24 and 72 hours (h) post surgery (PS)
Population: MITT; data from 1 site excluded due to GCP deviations
Measure: Number; unit: participants
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
participants
  24 h PS | 0 | 2 | 1 | 0
  72 h PS | 1 | 3 | 1 | 1
Statistical Analysis 1: Comparison: Pregabalin 150 mg vs Placebo; 24 h PS; Test type: Superiority or Other; p = 0.1927, Cochran-Mantel-Haenszel — P-values derived from CMH test adjusted for pooled centers. Centers with fewer than 8 treated subjests have been combined into pooled centers
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; 72 h PS; Test type: Superiority or Other; p = 0.3865, Cochran-Mantel-Haenszel — [p-value comment as in outcome 19, analysis 1]
Statistical Analysis 3: Comparison: Pregabalin 50 mg vs Placebo; 72 h PS; Test type: Superiority or Other; p = 0.9869, Cochran-Mantel-Haenszel — [p-value comment as in outcome 19, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin 150 mg vs Placebo; 72 h PS; Test type: Superiority or Other; p = 0.4354, Cochran-Mantel-Haenszel — [p-value comment as in outcome 19, analysis 1]
Statistical Analysis 5: Comparison: Pregabalin 300 mg vs Placebo; 72 h PS; Test type: Superiority or Other; p = 0.8061, Cochran-Mantel-Haenszel — [p-value comment as in outcome 19, analysis 1]

20. Secondary Outcome: Baseline and Change From Baseline in Anxiety Visual Analog Scale (VAS) Score
Description: Anxiety VAS is a single-item self-administered continuous measure of anxiety using a 100-millimeter (mm) line on which the subject is asked to place a mark indicating the intensity of current anxiety. The score is the distance in mm from the left-most point on the line to the subject's mark; range: 0 (Not at all anxious) at the left-most point to 100 (Extremely anxious) at the right-most point. Performed prior to blood draws.
Time Frame: Baseline; 2 hours (h) before surgery (BS); 1, 2, and 3 h PS; Days 2, 3, 4, 5, 6, 7, 8, and 9 PS
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on a scale
  Baseline (n=101, 98, 100, 100) | 20.2 (2.07) | 19.4 (2.10) | 18.4 (2.07) | 16.4 (2.07)
  2 h BS (n=101, 98, 100, 99) | 0.2 (1.56) | 3.2 (1.58) | 1.4 (1.54) | 4.2 (1.57)
  1 h PS (n=100, 96, 99, 99) | -6.4 (1.71) | -3.5 (1.73) | -5.2 (1.68) | -3.2 (1.70)
  2 h PS (n=101, 98, 100, 100) | -8.4 (1.51) | -7.6 (1.52) | -7.1 (1.48) | -6.1 (1.50)
  3 h PS (n=101, 98, 100, 100) | -8.7 (1.44) | -8.3 (1.45) | -9.0 (1.42) | -6.4 (1.43)
  Day 2 PS (n=101, 98, 100, 100) | -7.9 (1.59) | -10.4 (1.60) | -7.5 (1.56) | -5.8 (1.58)
  Day 3 PS (n=101, 97, 99, 100) | -9.1 (1.23) | -12.7 (1.25) | -11.3 (1.22) | -9.3 (1.23)
  Day 4 PS (n=101, 98, 98, 101) | -11.1 (1.23) | -15.3 (1.24) | -12.1 (1.23) | -11.4 (1.22)
  Day 5 PS (n=101, 98, 97, 99) | -12.3 (1.06) | -15.0 (1.07) | -12.4 (1.06) | -12.7 (1.07)
  Day 6 PS (n=100, 98, 97, 97) | -12.5 (1.08) | -15.0 (1.08) | -13.6 (1.07) | -12.8 (1.09)
  Day 7 PS (n=97, 93, 89, 95) | -13.0 (1.15) | -15.2 (1.16) | -13.3 (1.19) | -12.4 (1.15)
  Day 8 PS (n=61, 64, 53, 58) | -13.6 (1.16) | -15.4 (1.11) | -15.5 (1.25) | -14.7 (1.18)
  Day 9 PS (n=21, 24, 23, 22) | -16.6 (2.07) | -16.4 (1.90) | -14.7 (1.97) | -12.8 (1.90)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; Baseline; LS Means from ANOVA model with terms of treatment, pooled center, baseline VAS score and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.1682, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.2821, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.4781, ANOVA
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; 2 h BS; LS Means from ANOVA model with terms of treatment, pooled center, baseline VAS score and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0557, ANOVA
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 20, analysis 4]; Test type: Superiority or Other; p = 0.6098, ANOVA
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 20, analysis 4]; Test type: Superiority or Other; p = 0.1821, ANOVA
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; 1 h PS; LS Means from ANOVA model with terms of treatment, pooled center, baseline VAS score and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.1628, ANOVA
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 20, analysis 7]; Test type: Superiority or Other; p = 0.8999, ANOVA
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 20, analysis 7]; Test type: Superiority or Other; p = 0.3990, ANOVA
Statistical Analysis 10: Comparison: Pregabalin 50 mg vs Placebo; 2 h PS; LS Means from ANOVA model with terms of treatment, pooled center, baseline VAS score and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2665, ANOVA
Statistical Analysis 11: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 20, analysis 10]; Test type: Superiority or Other; p = 0.4885, ANOVA
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 20, analysis 10]; Test type: Superiority or Other; p = 0.6415, ANOVA
Statistical Analysis 13: Comparison: Pregabalin 50 mg vs Placebo; 3 h PS; LS Means from ANOVA model with terms of treatment, pooled center, baseline VAS score and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2269, ANOVA
Statistical Analysis 14: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 20, analysis 13]; Test type: Superiority or Other; p = 0.3228, ANOVA
Statistical Analysis 15: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 20, analysis 13]; Test type: Superiority or Other; p = 0.1808, ANOVA
Statistical Analysis 16: Comparison: Pregabalin 50 mg vs Placebo; Day 2 PS; LS Means from ANOVA model with terms of treatment, pooled center, baseline VAS score and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.3282, ANOVA
Statistical Analysis 17: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 20, analysis 16]; Test type: Superiority or Other; p = 0.0342, ANOVA
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 20, analysis 16]; Test type: Superiority or Other; p = 0.4198, ANOVA
Statistical Analysis 19: Comparison: Pregabalin 50 mg vs Placebo; Day 3 PS; LS Means from ANOVA model with terms of treatment, pooled center, baseline VAS score and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.9049, ANOVA
Statistical Analysis 20: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 20, analysis 19]; Test type: Superiority or Other; p = 0.0456, ANOVA
Statistical Analysis 21: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 20, analysis 19]; Test type: Superiority or Other; p = 0.2463, ANOVA
Statistical Analysis 22: Comparison: Pregabalin 50 mg vs Placebo; Day 4 PS; LS Means from ANOVA model with terms of treatment, pooled center, baseline VAS score and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.8231, ANOVA
Statistical Analysis 23: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 20, analysis 22]; Test type: Superiority or Other; p = 0.0221, ANOVA
Statistical Analysis 24: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 20, analysis 22]; Test type: Superiority or Other; p = 0.6974, ANOVA
Statistical Analysis 25: Comparison: Pregabalin 50 mg vs Placebo; Day 5 PS; LS Means from ANOVA model with terms of treatment, pooled center, baseline VAS score and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.7461, ANOVA
Statistical Analysis 26: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 20, analysis 25]; Test type: Superiority or Other; p = 0.1198, ANOVA
Statistical Analysis 27: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 20, analysis 25]; Test type: Superiority or Other; p = 0.8031, ANOVA
Statistical Analysis 28: Comparison: Pregabalin 50 mg vs Placebo; Day 6 PS; LS Means from ANOVA model with terms of treatment, pooled center, baseline VAS score and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.8515, ANOVA
Statistical Analysis 29: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 20, analysis 28]; Test type: Superiority or Other; p = 0.1285, ANOVA
Statistical Analysis 30: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 20, analysis 28]; Test type: Superiority or Other; p = 0.5561, ANOVA
Statistical Analysis 31: Comparison: Pregabalin 50 mg vs Placebo; Day 7 PS; LS Means from ANOVA model with terms of treatment, pooled center, baseline VAS score and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.6858, ANOVA
Statistical Analysis 32: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 20, analysis 31]; Test type: Superiority or Other; p = 0.0693, ANOVA
Statistical Analysis 33: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 20, analysis 31]; Test type: Superiority or Other; p = 0.5547, ANOVA
Statistical Analysis 34: Comparison: Pregabalin 50 mg vs Placebo; Day 8 PS; LS Means from ANOVA model with terms of treatment, pooled center, baseline VAS score and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.4610, ANOVA
Statistical Analysis 35: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 20, analysis 34]; Test type: Superiority or Other; p = 0.6640, ANOVA
Statistical Analysis 36: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 20, analysis 34]; Test type: Superiority or Other; p = 0.6158, ANOVA
Statistical Analysis 37: Comparison: Pregabalin 50 mg vs Placebo; Day 9 PS; LS Means from ANOVA model with terms of treatment, pooled center, baseline VAS score and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.1632, ANOVA
Statistical Analysis 38: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 20, analysis 37]; Test type: Superiority or Other; p = 0.1770, ANOVA
Statistical Analysis 39: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 20, analysis 37]; Test type: Superiority or Other; p = 0.4882, ANOVA

21. Secondary Outcome: Baseline and Change From Baseline in EuroQol (EQ-5D) Health State Profile Score
Description: EQ-5D is a self-administered questionnaire to assess health-related quality of life in 5 domains (mobility, self care, usual activities, pain or discomfort, and anxiety or depression). Scores from the 5 domains are used to calculate a single index value: the Health State Profile Score; range: 0.0 (death) to 1.0 (perfect health), higher scores indicating better health state.
Time Frame: Baseline and End of Treatment (EOT [Day 7 post surgery or Early Termination])
Population: MITT; data from 1 site excluded due to GCP deviations.
Measure: Least Squares Mean (Standard Error); unit: scores on scales
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on scales
  Baseline (n=101, 99, 100, 100) | 0.66 (0.015) | 0.68 (0.015) | 0.65 (0.015) | 0.66 (0.015)
  Change at EOT (n=97, 98, 99, 98) | -0.01 (0.016) | -0.01 (0.016) | -0.01 (0.015) | -0.04 (0.016)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; Baseline; LS Means from ANOVA model with terms of treatment, pooled center, baseline item score and basline PCS (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.7936, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.5092, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.4233, ANOVA
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; Change at EOT; LS Means from ANOVA model with terms of treatment, pooled center, baseline item score and basline PCS (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2033, ANOVA
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority or Other; p = 0.2142, ANOVA
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority or Other; p = 0.1218, ANOVA

22. Secondary Outcome: Change From Baseline in Pain Catastrophizing Scale (PCS) Total Score and Subscales
Description: The PCS is a self-administered questionnaire with 13 items, each scored from 0 (not at all) to 4 (all the time) for extent to which participant catastrophizes postoperative pain. Total score is sum of scores for all questions (range: 0 to 52); Subscale scores: Rumination (sum of scores for 4 items; range: 0 to 16); Magnification (sum of scores for 3 items; range: 0 to 12); and Helplessness (sum of scores for 6 items; range: 0 to 24); higher scores mean a greater extent of pain catastrophizing.
Time Frame: 3 hours (h) post surgery (PS) and End of Treatment (EOT [Day 7 PS or Early Termination])
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on a scale
  Total score change: 3 h PS (n=99, 98, 98, 99) | -3.5 (0.84) | -2.8 (0.85) | -3.6 (0.83) | -1.5 (0.84)
  Total score change: EOT (n=97, 96, 98, 96) | -6.2 (0.64) | -5.8 (0.64) | -6.3 (0.63) | -5.7 (0.64)
  Rumination change: 3 h PS (n=99, 98, 98, 99) | -1.0 (0.35) | -0.7 (0.35) | -1.1 (0.35) | -0.4 (0.35)
  Rumination change: EOT (n=97, 96, 98, 96) | -2.3 (0.28) | -1.8 (0.28) | -2.2 (0.27) | -1.9 (0.28)
  Magnification change: 3 h PS (n=99, 98, 99, 99) | -0.9 (0.21) | -0.9 (0.21) | -1.1 (0.21) | -0.7 (0.21)
  Magnification change: EOT (n=97, 96, 99, 96) | -1.5 (0.17) | -1.7 (0.17) | -1.6 (0.17) | -1.4 (0.17)
  Helplessness change: 3 h PS (n=99, 98, 99, 99) | -1.5 (0.37) | -1.3 (0.38) | -1.4 (0.37) | -0.5 (0.37)
  Helplessness change: EOT (n=97, 96, 99, 96) | -2.4 (0.27) | -2.3 (0.27) | -2.5 (0.26) | -2.5 (0.27)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; Total score change at 3 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0830, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Superiority or Other; p = 0.2339, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Superiority or Other; p = 0.0629, ANOVA
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; Total score change at EOT; LS Means from ANOVA model with terms of treatment, pooled center and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.5721, ANOVA
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Superiority or Other; p = 0.9713, ANOVA
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Superiority or Other; p = 0.4809, ANOVA
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; Rumination change at 3 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.1561, ANOVA
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 22, analysis 7]; Test type: Superiority or Other; p = 0.5267, ANOVA
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 22, analysis 7]; Test type: Superiority or Other; p = 0.1125, ANOVA
Statistical Analysis 10: Comparison: Pregabalin 50 mg vs Placebo; Rumination change at EOT; LS Means from ANOVA model with terms of treatment, pooled center and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.2965, ANOVA
Statistical Analysis 11: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 22, analysis 10]; Test type: Superiority or Other; p = 0.7774, ANOVA
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 22, analysis 10]; Test type: Superiority or Other; p = 0.3990, ANOVA
Statistical Analysis 13: Comparison: Pregabalin 50 mg vs Placebo; Magnification change at 3 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.4465, ANOVA
Statistical Analysis 14: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 22, analysis 13]; Test type: Superiority or Other; p = 0.4385, ANOVA
Statistical Analysis 15: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 22, analysis 13]; Test type: Superiority or Other; p = 0.2265, ANOVA
Statistical Analysis 16: Comparison: Pregabalin 50 mg vs Placebo; Magnification change at EOT; LS Means from ANOVA model with terms of treatment, pooled center and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.5985, ANOVA
Statistical Analysis 17: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 22, analysis 16]; Test type: Superiority or Other; p = 0.2146, ANOVA
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 22, analysis 16]; Test type: Superiority or Other; p = 0.3382, ANOVA
Statistical Analysis 19: Comparison: Pregabalin 50 mg vs Placebo; Helplessness change at 3 h PS; LS Means from ANOVA model with terms of treatment, pooled center and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.0430, ANOVA
Statistical Analysis 20: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 22, analysis 19]; Test type: Superiority or Other; p = 0.1128, ANOVA
Statistical Analysis 21: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 22, analysis 19]; Test type: Superiority or Other; p = 0.0632, ANOVA
Statistical Analysis 22: Comparison: Pregabalin 50 mg vs Placebo; Helplessness change at EOT; LS Means from ANOVA model with terms of treatment, pooled center and baseline PCS score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects were combined into pooled centers; Test type: Superiority or Other; p = 0.8667, ANOVA
Statistical Analysis 23: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 22, analysis 22]; Test type: Superiority or Other; p = 0.6365, ANOVA
Statistical Analysis 24: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 22, analysis 22]; Test type: Superiority or Other; p = 0.9275, ANOVA

23. Secondary Outcome: Relationship Between Baseline and Postoperative Pain Catastrophizing Scale (PCS) Score and Severity of Acute Pain and to Response to Therapy
Description: The PCS is a self-administered questionnaire with 13 items, each scored from 0 (not at all) to 4 (all the time) for extent to which participant catastrophizes postoperative pain. Total score is sum of scores for all items (range: 0 to 52); higher scores mean a greater extent of pain catastrophizing.
Time Frame: Baseline and Days 1 and 7 post surgery (PS)
Population: MITT; data from 1 site excluded due to GCP deviations. Data not analyzed as planned.
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

24. Secondary Outcome: Baseline and Change From Baseline in Short Form Acute Health Survey 12-Item Version (SF-12v2) Physical Component Summary Score (PCSS) and Mental Component Summary Score (MCSS)
Description: PCSS and MCSS are component summary scores from the self-administered SF-12v2 acute health quality of life, norm-based survey. PCSS range: 4.95 to 76.13; MCSS range: -0.79 to 79.69; lowest scores mean very much below and highest scores mean very much above the general population average.
Time Frame: Baseline and End of Treatment (EOT [Day 7 post surgery or Early Termination])
Population: MITT; data from 1 site excluded due to GCP deviations.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on a scale
  PCSS at baseline (n=101, 99, 100, 100) | 46.43 (0.914) | 48.14 (0.928) | 46.44 (0.915) | 44.89 (0.917)
  PCSS change at EOT (n=99, 99, 99, 98) | -6.86 (1.013) | -7.06 (1.021) | -6.92 (1.011) | -8.21 (1.025)
  MCSS at baseline (n=101, 99, 100, 100) | 54.48 (0.787) | 54.58 (0.799) | 54.81 (0.787) | 56.18 (0.789)
  MCSS change at EOT (n=99, 99, 99, 98) | 2.65 (0.764) | 2.68 (0.762) | 3.27 (0.750) | 1.50 (0.765)
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; PCSS at baseline; LS Means from ANOVA model with terms of treatment, pooled center and baseline score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects have were combined into pooled centers; Test type: Superiority or Other; p = 0.2136, ANOVA
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.0094, ANOVA
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.2131, ANOVA
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; PCSS change at EOT; LS Means from ANOVA model with terms of treatment, pooled center and baseline score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects have were combined into pooled centers; Test type: Superiority or Other; p = 0.3245, ANOVA
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 24, analysis 4]; Test type: Superiority or Other; p = 0.4070, ANOVA
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 24, analysis 4]; Test type: Superiority or Other; p = 0.3490, ANOVA
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; MCSS at baseline; LS Means from ANOVA model with terms of treatment, pooled center and baseline score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects have were combined into pooled centers; Test type: Superiority or Other; p = 0.1122, ANOVA
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 24, analysis 7]; Test type: Superiority or Other; p = 0.1380, ANOVA
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 24, analysis 7]; Test type: Superiority or Other; p = 0.2023, ANOVA
Statistical Analysis 10: Comparison: Pregabalin 50 mg vs Placebo; MCSS change at EOT; LS Means from ANOVA model with terms of treatment, pooled center and baseline score (for baseline visit ANOVA model with terms of treatment and pooled center). Centers with fewer than 8 treated subjects have were combined into pooled centers; Test type: Superiority or Other; p = 0.2639, ANOVA
Statistical Analysis 11: Comparison: Pregabalin 150 mg vs Placebo; [analysis description as in outcome 24, analysis 10]; Test type: Superiority or Other; p = 0.2524, ANOVA
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; [analysis description as in outcome 24, analysis 10]; Test type: Superiority or Other; p = 0.0832, ANOVA

25. Secondary Outcome: Participants With Chronic Postoperative Pain
Description: Number of participants who reported surgery-related pain at assessment (by answering 'yes' to a single question: "In the last 24 hours, have you had pain in the area affected by your surgery?")
Time Frame: 1, 3, and 6 months (mo) post surgery (PS)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
participants
  1 month PS (n=98, 98, 98, 99) | 20 | 24 | 19 | 26
  3 month PS (n=98, 97, 97, 97) | 3 | 5 | 5 | 3
  6 month PS (n=98, 97, 97, 97) | 1 | 1 | 1 | 0
Statistical Analysis 1: Comparison: Pregabalin 50 mg vs Placebo; 1 month PS; Test type: Superiority or Other; p = 0.2371, Cochran-Mantel-Haenszel — P-values are derived from Cochran-Mantel-Haenszel test adjusted for pooled centers. Centers with fewer than 8 treated subjects were combined into pooled centers
Statistical Analysis 2: Comparison: Pregabalin 150 mg vs Placebo; 1 month PS; Test type: Superiority or Other; p = 0.4435, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Pregabalin 300 mg vs Placebo; 1 month PS; Test type: Superiority or Other; p = 0.1692, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin 50 mg vs Placebo; 3 month PS; Test type: Superiority or Other; p = 0.8169, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Pregabalin 150 mg vs Placebo; 3 month PS; Test type: Superiority or Other; p = 0.5592, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; 3 month PS; Test type: Superiority or Other; p = 0.4453, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Pregabalin 50 mg vs Placebo; 6 month PS; Test type: Superiority or Other; p = 0.4795, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Pregabalin 150 mg vs Placebo; 6 month PS; Test type: Superiority or Other; p = 0.2733, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Pregabalin 300 mg vs Placebo; 6 month PS; Test type: Superiority or Other; p = 0.3173, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]

26. Secondary Outcome: Chronic Postoperative Pain: Pain Severity Index Score and Pain Interference Index Score on the Modified Brief Pain Inventory-Short Form (mBPI-sf)
Description: m-BPI-sf: a self-administered 11-point Likert rating scale to rate pain in the past 24 hours. Pain interference index score is mean of 7 individual item scores for interference of pain with functional activities (general activity, mood, walking ability, relations with other people, sleep, normal work, and enjoyment of life); range: 0 (does not interfere) to 10 (completely interferes with functional activities). Pain severity index score is mean of 4 individual item scores for pain severity (pain right now, and worst, least, and average pain); range: 0 (no pain) to 10 (worst imaginable pain).
Time Frame: 1, 3, and 6 months (mo) post surgery (PS)
Population: MITT; data from 1 site excluded due to GCP deviations; n=number of subjects who reported surgery-related pain at assessment (pregabalin 50 mg, pregabalin 150 mg, pregabalin 300 mg, and placebo, respectively). Data insufficient for standard deviation calculation at 6 mo PS.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on a scale
  Pain Severity 1 mo PS (n=20, 24, 19, 26) | 0.86 (0.801) | 0.81 (0.767) | 1.43 (1.210) | 0.76 (0.654)
  Pain Severity 3 mo PS (n=3, 5, 5, 3) | 0.58 (0.629) | 0.75 (0.354) | 1.55 (1.052) | 0.42 (0.520)
  Pain Interference 1 mo PS (n=20, 24, 19, 26) | 0.39 (0.630) | 0.71 (0.974) | 1.29 (1.463) | 0.51 (0.895)
  Pain Interference 3 mo PS (n=3, 5, 5, 3) | 0.14 (0.143) | 0.20 (0.163) | 1.34 (2.140) | 0.00 (0.000)

27. Secondary Outcome: Chronic Postoperative Pain: Total Score and Subscale Scores Using the Neuropathic Pain Symptom Inventory (NPSI)
Description: NPSI: a 12-item self-administered questionnaire to assess the characteristics of neuropathic pain on average in the last 24 hours. 5 subscale scores include: burning spontaneous (spont.) pain, pressing spont. pain, paroxysmal pain, evoked pain, and paresthesia or dysesthesia (paresth/dysesth) (range: 0 [no pain] to 10 [worst pain imaginable]); total score calculated from the 5 pain subscores (range: 0 to 0.5), higher scores meaning worse pain.
Time Frame: 1, 3, and 6 months (mo) post surgery (PS)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 102 | 99 | 101 | 101
scores on a scale
  NPSI total score 1 mo PS (n=20, 24, 19, 26) | 0.03 (0.025) | 0.03 (0.048) | 0.05 (0.038) | 0.04 (0.041)
  NPSI total score 3 mo PS (n=3, 5, 5, 3) | 0.02 (0.032) | 0.02 (0.022) | 0.05 (0.034) | 0.04 (0.044)
  Burning spont. pain 1 mo PS (n=20, 24, 19, 26) | 0.30 (0.571) | 1.04 (1.574) | 1.11 (1.761) | 0.77 (1.557)
  Burning spont. pain 3 mo PS (n=3, 5, 5, 3) | 1.00 (1.732) | 0.00 (0.00) | 0.40 (0.894) | 1.00 (1.732)
  Pressing spont. pain 1 mo PS (n=20, 24, 19, 26) | 0.43 (0.545) | 0.50 (1.189) | 1.03 (1.307) | 0.69 (0.939)
  Pressing spont. pain 3 mo PS (n=3, 5, 5, 3) | 0.50 (0.500) | 0.50 (0.354) | 2.30 (1.754) | 0.67 (0.764)
  Paroxysmal pain 1 mo PS (n=20, 24, 19, 26) | 0.95 (1.708) | 0.56 (1.106) | 1.05 (1.499) | 0.71 (1.133)
  Paroxysmal pain 3 mo PS (n=3, 5, 5, 3) | 0.33 (0.289) | 0.20 (0.274) | 0.70 (0.447) | 1.33 (1.528)
  Evoked pain 1 mo PS (n=20, 24, 19, 26) | 0.82 (0.970) | 0.76 (0.990) | 1.44 (1.495) | 1.05 (1.472)
  Evoked pain 3 mo PS (n=3, 5, 5, 3) | 0.22 (0.192) | 1.3 (2.082) | 1.73 (1.234) | 0.44 (0.509)
  Paresth/dysesth 1 mo PS (n=20, 24, 19, 26) | 0.10 (0.308) | 0.35 (0.961) | 0.32 (0.768) | 0.46 (0.774)
  Paresth/dysesth 3 mo PS (n=3, 5, 5, 3) | 0.50 (0.866) | 0.20 (0.274) | 0.10 (0.224) | 0.50 (0.866)

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) through post-treatment phone contact (Month 6)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin 50 mg | Pregabalin 150 mg | Pregabalin 300 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/108 | 1/106 | 0/103 | 3/108
Other Adverse Events (participants affected / at risk) | 46/108 | 44/106 | 56/103 | 45/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 50 mg (N=108) | Pregabalin 150 mg (N=106) | Pregabalin 300 mg (N=103) | Placebo (N=108)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 50 mg (N=108) | Pregabalin 150 mg (N=106) | Pregabalin 300 mg (N=103) | Placebo (N=108)
Bradycardia (Cardiac disorders) | 3 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 21 | 22 | 27 | 27
Nausea (Gastrointestinal disorders) | 21 | 18 | 14 | 22
Vomiting (Gastrointestinal disorders) | 2 | 7 | 1 | 6
Fatigue (General disorders) | 24 | 18 | 23 | 23
Pain (General disorders) | 1 | 0 | 3 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 3
Incision site pruritus (Injury, poisoning and procedural complications) | 0 | 1 | 4 | 3
Disturbance in attention (Nervous system disorders) | 11 | 11 | 15 | 16
Dizziness (Nervous system disorders) | 15 | 20 | 29 | 16
Headache (Nervous system disorders) | 5 | 3 | 1 | 3
Somnolence (Nervous system disorders) | 24 | 25 | 25 | 28
Confusional state (Psychiatric disorders) | 6 | 3 | 8 | 6
Insomnia (Psychiatric disorders) | 1 | 0 | 3 | 3
Dysuria (Renal and urinary disorders) | 10 | 6 | 10 | 10
Urinary retention (Renal and urinary disorders) | 1 | 3 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 7 | 4 | 6
Hypotension (Vascular disorders) | 7 | 3 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.